CLINICAL TRIAL: NCT06552520
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQH2722 Injection in the Treatment of Moderate to Severe Atopic Dermatitis in Subjects
Brief Title: To Evaluate the Phase III Clinical Trial of TQH2722 Injection in the Treatment of Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2722-III-01
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TQH2722 injection (Experimental): TQH2722 injection, 14 days for a treatment cycle
  Interventions: Drug: TQH2722 injection
- Placebo of TQH2722 injection (Placebo Comparator): Placebo of TQH2722 injection, 14 days for a treatment cycle
  Interventions: Drug: Placebo of TQH2722 injection

INTERVENTIONS:
Drug: TQH2722 injection — Humanized interleukin-4 receptor alpha (4Rα) monoclonal antibody
  Arms: TQH2722 injection
Drug: Placebo of TQH2722 injection — Placebo without drug substance
  Arms: Placebo of TQH2722 injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial with 500 participants. In this study, the safety evaluation used the common toxic reaction criteria of the National Cancer Institute to evaluate the adverse events of the drugs, and the effectiveness evaluation used the eczema area and severity score and the overall investigator score to confirm the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The age of signing the informed consent is 18-75 years old, regardless of gender.
* Meet the 2014 American Academy of Dermatology (AAD) standards, diagnosed as AD.
* During screening and baseline visit, eczema area and severity score (EASI) ≥16 points; Investigator global score (IGA) ≥3 points; Affected body surface area (BSA) ≥10%; Baseline pruritus Peak Value Scale (NRS) weekly mean ≥4 points.
* Have received at least 4 weeks of strong action or at least 2 weeks of super effective external glucocorticoid (TCS) treatment or sufficient duration of systemic glucocorticoid treatment, the efficacy is not sufficient; Or subjects cannot receive the above treatment due to adverse reactions or potential risks.

Exclusion Criteria:

* Used immunosuppressants/immunomodulatory drugs, ultraviolet phototherapy, systemic Chinese medicine treatment within 4 weeks before randomization.
* Received topical calcineurin inhibitors (TCS), topical calcineurin inhibitors (TCI), and other topical preparations within 2 weeks before randomization.
* Received anti-interleukin-4 receptor alpha (IL-4R) monoclonal antibodies, anti-ige monoclonal antibodies, or other biologic agents within 12 weeks or 5 half-lives (whichever is longer) prior to randomization.
* Had received live attenuated vaccine within 12 weeks prior to randomization or planned to receive it during the study period.
* Use of antihistamines within 1 week prior to randomization (unless you have received steady doses of antihistamines for at least 7 days).
* Received allergen specific immunotherapy within 6 months before randomization.
* There are skin comorbidities that may interfere with study evaluation.
* There is a history of clinically significant illness that the investigator believes poses a risk to the safety of the subject and is poorly controlled.
* A known or suspected history of immunosuppression (immune deficiency).
* Subjects with any type of active malignancy or a history of malignancy (except cervical cancer or non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma, and papillary thyroid carcinoma that have been cured for more than 5 years prior to the screening period).
* Subject may have active Mycobacterium tuberculosis infection.
* Subjects with severe liver and kidney function impairment.
* Screening period HIV antibody positive, or have a history of HIV infection.
* Screening period of treponema pallidum antibody positive.
* Participated in clinical trials of other drugs or medical devices within 12 weeks prior to randomization.
* Treatment-requiring infections were present in the 4 weeks prior to randomization.
* During the study period, subjects plan to undergo major surgical operations.
* Pregnant or lactating women.
* Alcohol, drug abuse and known drug dependence.
* History of atopic keratoconjunctivitis with corneal involvement.
* The subject has any medical or psychiatric symptoms that interfere with participation in the study or with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Participants who achieved EASI-75 (≥75% improvement from baseline) on the eczema Area and Severity score (EASI) | Baseline to 16 weeks after treatment
  Percentage of participants who achieved EASI-75 (≥75% improvement from baseline) on the eczema Area and Severity score (EASI)
Subjects with an Investigator's Overall Rating (IGA) score (5-scale) of 0 or 1 and ≥2 points decline from baseline | Baseline to 16 weeks after treatment
  Percentage of subjects with an Investigator's Overall Rating (IGA) score (5-scale) of 0 or 1 and ≥2 points decline from baseline.

SECONDARY OUTCOMES:
The incidence of adverse events | After medication to 60 weeks
  Adverse events that occur during treatment
Steady valley concentration of TQH2722 | After medication to 60 weeks
  Relatively stable concentration levels of TQH2722
The incidence and titer of drug-resistant antibodies (ADA) in subjects | After medication to 60 weeks
  The incidence and titer of drug-resistant antibodies (ADA) in subjects
Incidence of neutralizing antibodies (Nab) | After medication to 60 weeks
  Incidence of neutralizing antibodies (Nab)
Eczema area and severity score (EASI) change from baseline | From baseline to week 60
  The affected area of each site was assessed. According to the percentage of the affected area, the corresponding Region score was 0 to 6. The higher the score, the more severe the involvement.
Rate of change from baseline in the Investigator's overall Score (IGA) | After medication to 60 weeks
  The researchers assessed the form of the dermatitis using a 5-point scale (0-5), with higher scores being more severe.
Change of body surface area from baseline in moderate to severe atopic dermatitis | After medication to 60 weeks
  The researchers used a nine-point scale to assess the percentage of AD affected area in the whole body (0-100%), with the larger the value, the more severe the involvement.
Change rate of atopic dermatitis score (SCORAD) from baseline | After medication to 60 weeks
  According to the involvement of skin surface area, the severity of skin lesions and the subjective symptom score, the higher the value, the more severe the dermatitis.
Change in daily Peak Itch Digital Rating Scale (NRS) score from baseline | After medication to 60 weeks
  Rate the most severe itching in the past 24 hours on a scale of 0-10, with higher numbers being more severe.
Rate of change in dermatological quality of life (DLQI) score from baseline | After medication to 60 weeks
  Assess how much the skin problems of the last week have affected the subjects' lives
Change in patients' self-assessment of eczema (POEM) from baseline | After medication to 60 weeks
  The number of days in the past 7 days to assess whether eczema caused skin problems such as itching and bleeding, 0 indicates no days, 1 indicates 1-2 days, 2 indicates 3-4 days, 3 indicates 5-6 days, and 4 indicates all days.

CONTACTS AND LOCATIONS:
Locations (72):
- China (72):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Tongling People's Hospital, Tongling, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of the Chinese People's Liberation Army Army Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Medical College affiliated People's Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Dermatology Hospital of Southern Medical UniversityDermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Qiqihar Hospital of Traditional Chinese Medicine, Qiqihar, Heilongjiang
  - Anyang District Hospital, Puyang City, Anyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang city first People's Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Xiangya Third Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Hunan Medical University General Hospital, Huaihua, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Second Hospital of Jilin University, Changchun, Jilin
  - Panjin Liao oil precious stone flower hospital, Panjin, Liaoning
  - Yinchuan First People's Hospital, Yinchuan, Ningxia
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Dezhou People's Hospital, Dezhou, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Peking University First Hospital Taiyuan Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of PLA Air Force Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi 'an Medical College, Xi’an, Shanxi
  - The Second Affiliated Hospital of the Chinese People's Liberation Army Air Force Medical University, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Jiaxing second Hospital, Jiaxing, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang